CLINICAL TRIAL: NCT04276844
Title: Incidence of Postoperative Persistent Diaphragmatic Dysfunctions in Cardiac Surgery
Acronym: INDYD
Status: Completed | Type: Observational
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Other Study IDs: 2019/06
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Surgery, Cardiac
Keywords: Diaphragmatic paralysis; Respiratory complications
MeSH Terms: conditions — Respiratory Paralysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non diaphragmatic dysfunction at day 7 post-surgery: Diaphragmatic displacement after sniff test ≥ 16 mm for women and ≥ 18 mm for men
  Interventions: Diagnostic Test: Ultrasonography using the two-dimensional (2D) mode
- Persistent diaphragmatic dysfunction at day 7 post-surgery: Diaphragmatic displacement after sniff test < 16 mm for women and < 18 mm for men
  Interventions: Diagnostic Test: Ultrasonography using the two-dimensional (2D) mode; Diagnostic Test: Respiratory Functional Explorations

INTERVENTIONS:
Diagnostic Test: Ultrasonography using the two-dimensional (2D) mode — Diaphragmatic amplitude assessed by ultrasonography during quiet breathing and after sniff test, before the surgery and at day 7 post-surgery in all patients.
Diagnostic Test: Respiratory Functional Explorations — Forced vital capacity (FVC), forced expiratory volume in 1 second (FEV) and total lung capacity (TLC) measured at day 7
  Groups: Persistent diaphragmatic dysfunction at day 7 post-surgery

SUMMARY:
Postoperative respiratory complication is a common complication that occurs in 6% of patients after cardiac surgery and increases morbidity and mortality and hospital length of stay. Diaphragmatic dysfunction (DD) is one of the main risk factors for post-operative respiratory distress syndrome. It alters the ventilatory mechanical function of patients and promotes pneumonia. In the literature, risk factors included older age, diabetes, harvesting of a mammary artery, intraoperative ice solution using, prolonged cardiopulmonary bypass and intra-operative phrenic nerve injury.

Ultrasonography using the two-dimensional (2D) mode is a diagnosis tool for DD. For patients with DD, ultrasound criteria are: 1) an excursion during quiet breathing < 9 mm for woman and < 10 mm for man, 2) an excursion after sniff test < 16 mm for woman and < 18 mm for man and 3) an excursion during deep breathing < 37 mm for woman and < 47 mm for man. A paradoxical diaphragmatic ascent may also be observed during inspiration.

DD may be transient, linked to mechanical factors such as pain, the presence of pleural and mediastinal drains, lying down or sternotomy; with recovery from 5 postoperative days. It may be more prolonged (persistent after 7 days) in connection with a partial or complete phrenic nerve injury and / or diaphragmatic devascularization after mammary artery harvesting.

The aim of this prospective study is to determine the incidence of persistent DD after cardiac surgery.

DETAILED DESCRIPTION:
Diaphragmatic amplitude will be assessed by ultrasonography during quiet breathing and after sniff test, before the surgery and at day 7 post-surgery in all patients.

Patients with persistent DD at day 7 post-surgery will have additional Respiratory Functional Explorations.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery requiring sternotomy
* Consent for participation
* Affiliation to the social security system

Exclusion Criteria:

* Contraindication to preoperative respiratory functional explorations
* Pregnant or breastfeeding women
* Patients under protection of the adults (guardianship, curators or safeguard of justice)
* Communication difficulties or neuropsychiatric disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 150 patients undergoing cardiac surgery
Sampling Method: Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Incidence of persistent diaphragmatic dysfunctions after cardiac surgery | 8 days
  Diaphragmatic excursion measured during sniff test (displacement, mm)

SECONDARY OUTCOMES:
Incidence of respiratory complications | up to 2 months
  Occurrence of pneumonia, atelectasis requiring bronchial clearing by fibroscopy, reintubation, prolonged mechanical ventilation (>24h) or prolonged non-invasive ventilation (>48h)
Intensive Care Unit (ICU) length of stay | up to 2 months
  Duration of ICU stay measured in days
Hospital length of stay | up to 2 months
  Duration of hospitalization measured in days
Respiratory function test in the group with persistent diaphragmatic dysfunction | 8 days
  Forced vital capacity (FVC), forced expiratory volume in 1 second (FEV) and total lung capacity (TLC) measured at day 7 and compared to day 0

CONTACTS AND LOCATIONS:
Locations (1):
- CMC Ambroise Paré, Neuilly-sur-Seine, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Laghlam D, Naudin C, Srour A, Monsonego R, Malvy J, Rahoual G, Squara P, Nguyen LS, Estagnasie P. Persistent diaphragm dysfunction after cardiac surgery is associated with adverse respiratory outcomes: a prospective observational ultrasound study. Can J Anaesth. 2023 Feb;70(2):228-236. doi: 10.1007/s12630-022-02360-8. Epub 2022 Dec 13. PMID 36513852